CLINICAL TRIAL: NCT06110832
Title: The Effect of Mindfulness-based Yoga and Meditation Practices on Stress, Self-esteem, Body Image and Sexual Adjustment in Breast Cancer Patients Undergoing Modified Radical Mastectomy: A Randomized Controlled Trial
Brief Title: The Effect of Mindfulness-based Yoga and Meditation on Some Parameters in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Collaborators: Koç University (Other)
Responsible Party: Principal Investigator, Melike Pehlivan, Lecturer, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KHSU-GSHMYO-MP-01
Record Dates: First submitted 2023-10-23; First posted 2023-11-01 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
Keywords: stress; body image; self esteem; sexual desire
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: 2-arm study with experimental control groups
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the research, the researcher is involved in the implementation of the mindfulness-based meditation and yoga program, data collection and data entry into the system. At the same time, the women in the experimental group had to be informed about the research. Therefore, researcher and participant blinding could not be performed. The data obtained from the research were coded as Group 1 and Group 2 by the researcher and transferred to the analysis program. The statistical expert who performed the analysis had no knowledge about the groups. Thus, it was aimed to control statistical bias, control bias and detection bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based Meditation and Yoga Intervention Group (Experimental): After randomization, participants in the experimental group underwent mindfulness-based meditation and yoga practices with 90-minute sessions on Thursdays for 8 weeks. In these practices, a different theme was determined each week.
  The 8-week theme headings are as follows:
  Week 1 exploring mindfulness Week 2: How do we perceive the world? week 3 being in the body Week 4 meeting stress with mindful awareness Week 5 our relationship with stress-inducing thoughts Week 6 Communication with mindfulness Week 7 taking care of yourself Week 8 farewell and a new beginning
  Interventions: Behavioral: Mindfulness-based Meditation and Yoga program
- Control Group (No Intervention): No intervention was applied to the control group

INTERVENTIONS:
Behavioral: Mindfulness-based Meditation and Yoga program — In the mindfulness-based meditation and yoga program, mindfulness-based formal and informal interventions are conducted for 8 weeks.
  Arms: Mindfulness-based Meditation and Yoga Intervention Group

SUMMARY:
The purpose of this study was to evaluate the effect of mindfulness-based meditation and yoga on stress, self-esteem, body image and sexual adjustment in breast cancer patients.

DETAILED DESCRIPTION:
The study was conducted in a single-center, prospective (pretest-posttest-2. month follow-up), two-arm (1:1), randomized controlled experimental design.

In this study, the effects of an 8-week structured mindfulness-based meditation and yoga program on stress, self-esteem, body image and sexual adjustment will be evaluated in women undergoing modified radical mastectomy. The 8-week interventions were conducted by the researcher. The researcher who performed these applications has a certificate of mindfulness meditation, yoga, breathing and movement trainer. Due to the nature of the research, the researcher is involved in the implementation of the mindfulness-based meditation and yoga program, data collection and data entry into the system. At the same time, the women in the experimental group had to be informed about the research. Therefore, researcher and participant blinding could not be performed. However, randomization was performed to prevent selection bias (1:1). The randomization process was performed by a statistical expert other than the researcher and communicated to the researcher. The participants included in the study were numbered from 1 to 41, preserving their random order in the list received from the hospital. The groups were divided into Group 1 and Group 2 by the statistician and the first group was determined as the experimental group and the second group as the control group by lottery method. The randomization table was created by making use of "http://calculatorsoup.com". Before the 8-week process started, 3 measurements were made to the participants: pre-test, post-test at the end of 8 weeks and follow-up measurement 2 months after the application.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and write Turkish,
* Who have undergone modified radical mastectomy surgery,
* Female patients between the ages of 30-55,
* Premenopausal patients,
* At least 3 months have passed since the mastectomy operation and all available treatments (chemotherapy and/or radiotherapy treatments),
* No condition that constitutes an obstacle for active sexual life (for sexual compatibility assessment),
* Those who have not undergone plastic and reconstructive surgery for the breast after modified radical mastectomy,
* Those who have no previous meditation and/or yoga experience,
* Those who do not have a diagnosis of a mental disorder of organic origin,
* Those who do not have substance and/or alcohol addiction,
* Those who do not have severe depression accompanying the disease,
* Those who do not have a physical disability that would prevent participation in the study,
* Those who agree to participate in the study will be included in the sample.

Exclusion Criteria:

* Patients who received neoadjuvant chemotherapy in the preoperative period,
* Patients under the age of 30 and over the age of 55,
* Patients who have undergone oncoplastic, breast-conserving surgery,
* Patients with previous experience of mindfulness, meditation or yoga will not be included in the study.

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2023-05-11 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale | Week 1 (pre-test), Week 8 (final test) and 2nd month (follow-up measurement)
  The Perceived Stress Scale developed by Cohen, Kamarck and Mermelstein (1983) consists of 14 items and has 2 sub-dimensions (perception of inadequate self-efficacy and perception of stress/discomfort). Individuals are asked to rate on a 5-point Likert scale how often they have experienced certain feelings or thoughts in the last month.

SECONDARY OUTCOMES:
Rosenberg Self-Esteem Scale | Week 1 (pre-test), Week 8 (final test) and 2nd month (follow-up measurement)
  Rosenberg Self-Esteem Scale is a self-report scale consisting of 63 multiple-choice questions. The scale consists of twelve subcategories. Rosenberg stated that the subscales can be used separately in research if desired. For the purpose of the study, the first '10' items of the scale will be used to measure self-esteem.
Sexual Compliance and Body Image Scale | Week 1 (pre-test), Week 8 (final test) and 2nd month (follow-up measurement)
  The scale was developed by Dalton et al. to assess body image and sexuality in postoperative women with breast cancer. It consists of two separate scales, the Body Image Scale and the Sexual Adjustment Scale. The six-item Body Image Scale has two subscales, namely before body image score and after body image score. These subscales measure body image before and after breast cancer diagnosis. The eight-item Sexual Adjustment Scale has three subscales: sexual adjustment, sexual functioning and sexual importance of breasts score.
Female Sexual Function Scale | Week 1 (pre-test), Week 8 (final test) and 2nd month (follow-up measurement)
  It is a personal tool for measuring sexual function that has been validated in women who have been clinically diagnosed with female sexual dysfunction. The Female Sexual Function Scale was developed by Rosen et al. in the USA in 2000 as a 19-item multidimensional scale to assess female sexual function.

CONTACTS AND LOCATIONS:
Overall Officials: Melike Pehlivan, Principal Investigator — Kutahya Health Science University; Semra Eyi, Study Director — Osmangazi University
Locations (1):
- Kutahya Health Science University, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pehlivan M, Eyi S. The Impact of Mindfulness-Based Meditation and Yoga on Stress, Body Image, Self-esteem, and Sexual Adjustment in Breast Cancer Patients Undergoing Modified Radical Mastectomy: A Randomized Controlled Trial. Cancer Nurs. 2025 May-Jun 01;48(3):190-199. doi: 10.1097/NCC.0000000000001427. Epub 2024 Nov 18. PMID 39773822